CLINICAL TRIAL: NCT00566215
Title: Clinical and Hormonal Study of a New Surgical Treatment of Type 2 Diabetes Mellitus: Duodenal Exclusion Associated With Omentectomy
Brief Title: Treatment of Type 2 Diabetes Mellitus by Duodenal Exclusion Associated With Omentectomy: Clinical and Hormonal Study
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Benefit of duodenal exclusion alone less than expected for treatment of type 2 diabetes; an additional effect of combination with omentectomy not observed
Sponsor: University of Campinas, Brazil (Other)
Responsible Party: Bruno Geloneze, University of Campinas, Brazil
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LIMED0003
Record Dates: First submitted 2007-11-30; First posted 2007-12-03 (Estimated); Last update posted 2010-07-23 (Estimated); Status verified 2010-07

CONDITIONS: Diabetes Mellitus, Type 2; Insulin Resistance; Obesity
Keywords: diabetes mellitus, type 2; Insulin resistance; Intra-Abdominal Fat; Omentum; duodenal exclusion; bariatric surgery; Glucagon-Like Peptide 1; Gastric Inhibitory Polypeptide; insulin; glucagon; ghrelin; adiponectin; Cytokines
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Insulin Resistance; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Duodenal exclusion plus total omentectomy
  Interventions: Procedure: Duodenal exclusion plus omentectomy
- 2 (Active Comparator): Duodenal exclusion without omentectomy
  Interventions: Procedure: Duodenal exclusion without omentectomy

INTERVENTIONS:
Procedure: Duodenal exclusion plus omentectomy — Under open laparotomy, a duodenum section 2cm below the pylorus and a jejunum section below Treitz's Angle to create a excluded biliopancreatic limb of 150cm. A Roux-in-Y retrocolic anastomosis of the alimentary limb promotes the gastrojejunal continuity and the anastomosis of the excluded biliopancreatic limb is done 100cm below the jejunal-pyloric union.
  Additionally, total omentectomy is performed.
  Other Names: Duodenojejunal exclusion plus omentectomy; Duodenal-jejunal bypass plus omentectomy
  Arms: 1
Procedure: Duodenal exclusion without omentectomy — Under open laparotomy, a duodenum section 2cm below the pylorus and a jejunum section below Treitz's Angle to create a excluded biliopancreatic limb of 150cm. A Roux-in-Y retrocolic anastomosis of the alimentary limb promotes the gastrojejunal continuity and the anastomosis of the excluded biliopancreatic limb is done 100cm below the jejunal-pyloric union.
  Other Names: Duodenojejunal exclusion; Duodenal-jejunal bypass
  Arms: 2

SUMMARY:
Based in a surgery technique studied in a non-obese diabetic mouse model by Rubino and Marescaux(2004), wich reversed diabetes in those animals, we have performed a previous study in human volunteers with type 2 diabetes and overweight (non-obese). The surgery is a duodenal exclusion in wich the stomach volume is kept intact. We observed improvement of glycemic control and hemoglobin A1c, allied to reduction of medicines: insulin was withdrawn or significantly lowered.

Further improvement of diabetes could be achieved by intervention in insulin resistance, another factor of diabetes pathophysiology. As that factor is related to visceral fat, we hypothesize that surgical removal of the major omentum, a great component of central adiposity, could beneficial .

This study will evaluate the mechanisms of amelioration of type 2 diabetes mellitus after duodenal exclusion surgery plus total omentectomy, by the method of standardized meal stimulus and insulin tolerance test, in human non-obese volunteers with diabetes type 2 and known insulin secretion capacity.

The previously studied volunteers submitted to duodenal exclusion without omentectomy will be the control group.

DETAILED DESCRIPTION:
Diabetes reversion is observed after bariatric surgeries even before significant weight loss could explain it, mainly in predominantly malabsorptive procedures, followed by those combining malabsorption and gastric restriction. Changes in the hormonal communication between the digestive system (incretins)and the pancreas would explain the antidiabetogenic role of the surgery, so this effect could be obtained in nonobese, diabetic individuals.

Based in a surgery technique studied in a non-obese diabetic mouse model by Rubino and Marescaux(2004), wich reversed diabetes in those animals, we have performed a previous study in human volunteers with type 2 diabetes and overweight (non-obese). The surgery is a duodenal exclusion: the stomach volume is kept intact, maintaining the caloric ingestion and the weight reduces less than 5%, without the potential nutritional deprivations commonly seen in the bariatric surgery. We observed improvement of glycemic control and hemoglobin A1c, allied to reduction of medicines: insulin was withdrawn or significantly lowered. An standardized mixed meal tolerance test showed favorable changes in the gastrointestinal hormones that stimulate insulin secretion (incretins): increase of GLP-1 and reduction of GIP.

Further improvement of diabetes could be achieved by intervention in insulin resistance, another factor of diabetes pathophysiology. As that factor is related to visceral fat, we hypothesize that surgical removal of the major omentum, a great component of central adiposity, could beneficial .

In fact, surgical removal of visceral fat in rodents improves insulin sensitivity. A pilot study in human, obese volunteers submitted to gastric adjustable band was promising int this aspect.

This study will evaluate the mechanisms of amelioration of type 2 diabetes mellitus after duodenal exclusion surgery plus total omentectomy , by the method of standardized meal stimulus and insulin tolerance test, in human non-obese, volunteers with diabetes type 2 and known insulin secretion capacity.

The previously studied volunteers submitted to duodenal exclusion without omentectomy will be the control group.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 to 60 years.
* BMI between 25 and 29,9 kg/m².
* Weight variance less than 5% in the last 3 months.
* Previous diagnosis of diabetes type 2.
* Insulin requirement, alone or along with oral agents
* Capacity to understand the procedures of the study.
* To agree voluntarily to participate of the study, signing an informed consent.

Exclusion Criteria:

* Positive Anti-GAD antibodies
* Laboratorial signal of probable failure of insulin production, i. e., seric peptide C lesser than 1 ng/mL.
* History of hepatic disease like cirrhosis or chronic active hepatitis.
* Kidney dysfunction (creatinine > 1,4 mg/dl in women and > 1,5 mg/dl in men).
* Hepatic dysfunction: ALT and/or AST 3x above upper normal limit.
* Recent history of neoplasia (< 5 years).
* Use of oral or injectable corticosteroids for more than consecutive 14 days in the last three months.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2007-07; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Improvement or reversal of type 2 diabetes mellitus | 7 days, 14 days, 21 days, 1 month, 2 months, 3 months, six months and one year

SECONDARY OUTCOMES:
Changes in the secretion pattern of incretins, insulin and glucagon after intervention, as measured by standardized mixed meal tolerance test | 2 months, 6 months and 1 year
Changes in body weight and fat distribution after intervention | 1 month, 2 months, 3 months, 6 months and 1 year
Changes in seric free fatty acids and lipoproteins | one month, 2 months, 3 months, 6 months and 1 year
Regression of carotid intima-media thickness | 1 month, 3 months, 6 months and 1 year
Changes in seric levels of adiponectin and other adipokines. | 2 months, 6 months and 1 year
Improvement of insulin sensitivity as measured by insulin tolerance test. | 1 month, 3 months, 6 months and 1 year

CONTACTS AND LOCATIONS:
Overall Officials: José Carlos Pareja, MD, PhD, Principal Investigator — University of Campinas (UNICAMP); Bruno Geloneze, MD, PhD, Principal Investigator — University of Campinas (UNICAMP)
Locations (1):
- LIMED (Laboratory of Investigation of Metabolism and Diabetes)/GASTROCENTRO/Univeristy of Campinas (UNICAMP), Campinas, São Paulo, Brazil

REFERENCES:
- [Background] Rubino F, Marescaux J. Effect of duodenal-jejunal exclusion in a non-obese animal model of type 2 diabetes: a new perspective for an old disease. Ann Surg. 2004 Jan;239(1):1-11. doi: 10.1097/01.sla.0000102989.54824.fc. PMID 14685093
- [Background] Thorne A, Lonnqvist F, Apelman J, Hellers G, Arner P. A pilot study of long-term effects of a novel obesity treatment: omentectomy in connection with adjustable gastric banding. Int J Obes Relat Metab Disord. 2002 Feb;26(2):193-9. doi: 10.1038/sj.ijo.0801871. PMID 11850750
- [Background] Pitombo C, Araujo EP, De Souza CT, Pareja JC, Geloneze B, Velloso LA. Amelioration of diet-induced diabetes mellitus by removal of visceral fat. J Endocrinol. 2006 Dec;191(3):699-706. doi: 10.1677/joe.1.07069. PMID 17170226
- [Background] Barzilai N, She L, Liu BQ, Vuguin P, Cohen P, Wang J, Rossetti L. Surgical removal of visceral fat reverses hepatic insulin resistance. Diabetes. 1999 Jan;48(1):94-8. doi: 10.2337/diabetes.48.1.94. PMID 9892227
- [Background] Gabriely I, Ma XH, Yang XM, Atzmon G, Rajala MW, Berg AH, Scherer P, Rossetti L, Barzilai N. Removal of visceral fat prevents insulin resistance and glucose intolerance of aging: an adipokine-mediated process? Diabetes. 2002 Oct;51(10):2951-8. doi: 10.2337/diabetes.51.10.2951. PMID 12351432
- [Result] Geloneze B, Geloneze SR, Fiori C, Stabe C, Tambascia MA, Chaim EA, Astiarraga BD, Pareja JC. Surgery for nonobese type 2 diabetic patients: an interventional study with duodenal-jejunal exclusion. Obes Surg. 2009 Aug;19(8):1077-83. doi: 10.1007/s11695-009-9844-4. Epub 2009 May 12. PMID 19475464